CLINICAL TRIAL: NCT00603928
Title: Placebo Interventions in General Practice
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Academy of Medical Sciences (SAMS) (Other)
Responsible Party: Nikola Biller-Andorno, University of Zurich, Institute for Biomedical Ethics
Other Study IDs: RRMA-5-07
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: General Practitioners
Keywords: attitude; attitude of health personnel; ethics; bioethics; biomedical ethics; patient care; physicians; placebo effect; placebos; questionnaires; therapy; general practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Physicians often have an ambivalent relationship to placebo interventions. On the one hand they know of the intriguing effect of sugar pills or saline infusions but on the other hand they mostly feel constrained to adopt scientifically proven, specific therapies for ethical reasons. Against the background of international literature one can assume that also Swiss general practitioners use several forms of placebo interventions in a significant part of their patients.

The aim of the project is to ascertain to which extent and in which way Swiss general practitioners make use of placebo interventions. Furthermore knowledge of the mode of action of placebo interventions and the perceived moral and lawful permissibility of placebo interventions and the presumed attitudes of the patients will be investigated.

The empicical core of the study is a questionnaire survey of general practitioners in urban and rural areas of Switzerland. The results and conclusions of the survey will be discussed during a workshop with interested GPs, researchers and ethicists.

The obtained data will lead to a better understanding of the application of placebo interventions in the general practice in Switzerland (how often and in which manner, accompanied by what information, for which diseases and for which patient groups placebos are applied). Moreover the study will help to articulate potential moral ambiguities of physicians using placebo interventions.

ELIGIBILITY:
Inclusion Criteria:

* general practitioners and pediatricians in medical practice of the canton Zurich in Switzerland

Exclusion Criteria:

* no patient encounters

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: general practitioners and pediatricians in medical practice of the canton Zurich in Switzerland
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland